CLINICAL TRIAL: NCT00338221
Title: Prospective Double Blinded Randomized Clinical Trial of Alanyl-Glutamine or Glycine in Children With Persistent Diarrhea or Malnutrition
Brief Title: Clinical Trial of Alanyl-Glutamine or Glycine in Children With Persistent Diarrhea or Malnutrition
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Richard L. Guerrant, MD, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02-039
Record Dates: First submitted 2006-06-15; First posted 2006-06-20 (Estimated); Last update posted 2008-10-28 (Estimated); Status verified 2008-10

CONDITIONS: Diarrhea, Malnutrition
Keywords: Diarrhea, Malnutrition, Brazil
MeSH Terms: conditions — Diarrhea; Malnutrition | interventions — alanylglutamine; Glycine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: alanyl-glutamine
Drug: glycine

SUMMARY:
This is a double blinded randomized clinical trial of Alanyl-Glutamine or Glycine in children with persistent diarrhea or malnutrition. The primary objective of the study is to determine the effect of 7 days of supplementation of alanyl-glutamine as it compares to glycine on the damaged intestinal barrier function, measured by lactulose/mannitol test on day 8, in children at HIAS in Fortaleza, Ce, Brazil, with persistent diarrhea (history > 2 weeks duration) or malnutrition.

DETAILED DESCRIPTION:
This is a double blinded randomized clinical trial of Alanyl-Glutamine or Glycine in children with persistent diarrhea or malnutrition. The primary objective of the study is to determine the effect of 7 days of supplementation of alanyl-glutamine as it compares to glycine on the damaged intestinal barrier function, measured by lactulose/mannitol test on day 8, in children at HIAS in Fortaleza, Ce, Brazil, with persistent diarrhea (history > 2 weeks duration) or malnutrition (assessed by height-for-age Z-score less than -1). Secondary objectives of the study include determining the effect of 7 days of supplementation of alanyl-glutamine or glycine on diarrhea frequency and duration; weight gain; protein loss and intestinal inflammation, and lactoferrin excretion; and weight gain at 2-4 weeks after treatment. One hundred and eight children who meet the inclusion criteria will be prospectively randomized to one of two treatment groups: (1) Glycine or (2) Alanyl-Glutamine. All children will be given vitamin A and Zinc supplementation; and if they have diarrhea, standard oral or IV rehydration therapy will be administered.

ELIGIBILITY:
Inclusion Criteria:

1. Children ages 3 to 36 months with a history of persistent diarrhea (3 or more unformed stools/day) for > 2 weeks or height-for-age Z-score (HAZ) less than -1, which is the median of HAZ scores in children at HIAS.
2. Be an inpatient and willing to stay for 7 nights at HIAS.
3. Child's parent or guardian must sign informed consent.

Exclusion Criteria:

1. Children exclusively breast-fed (Reason: The diet needs to be controlled in order to evaluate the study treatment effect)
2. Children who participated in the "community study" or any other study within the past two years (Reason: The children in the "community study" will have received glutamine.)
3. Children with suspected other illnesses as indicated by fever >102 degrees F at time of screening off antipyretics.
4. Children with suspected systemic disease at the time of screening including but not limited to shock, meningitis, sepsis, pneumonia, tuberculosis, varicella
5. Severe malnutrition defined as HAZ <-3.

Ages: 3 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108
Dates: Start 2004-08; Study Completion 2005-04

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Guerrrant, MD, Principal Investigator — University of Virginia